CLINICAL TRIAL: NCT01316354
Title: Effect of Arabinoxylan and Beta-glucan Compared With Whole Grain and Whole Meal Bread in Subjects With the Metabolic Syndrome
Brief Title: Effect of Dietary Fibre and Whole Grain on the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, AnneMarie Kruse, Professor Kjeld Hermansen, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-BioFunCarb
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Metabolic Syndrome
Keywords: Arabinoxylan; Beta glucan; Whole grain; Dietary fibre; Metabolic syndrome; Glycemic index; Satiety
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Beta-glucan (Experimental): Bread with purified beta-glucan
  Interventions: Other: Bread types
- Rye kernels (Experimental): Rye bread with kernels
  Interventions: Other: Bread types
- White bread (Experimental): White bread
  Interventions: Other: Bread types
- Arabinoxylan (Experimental): Bread with Purified arabinoxylan
  Interventions: Other: Bread types

INTERVENTIONS:
Other: Bread types — Bread with 50 g available carbohydrate

SUMMARY:
Sedentary lifestyles and increasing obesity are main causes of the global increase in the prevalence of the metabolic syndrome (Mets) and type 2 diabetic (T2DM). Diet quality, particularly composition of carbohydrate play also a significant role. The glycemic index (GI) describes in relative terms rise of blood glucose after ingestion of carbohydrate-rich food. Purified dietary fibre as β-glucan (BG) has been shown to reduce GI and affect levels of satiety hormones. In contrast, our knowledge of the physiological effects of arabinoxylans (AX), which constitute a substantial part of dietary fibre in cereal products, is limited. The investigators also lack a deeper understanding of the importance of whole grain (whole grain with whole kernels, and purified dietary fibre) in relation to Mets and T2DM.

Hypothesis: The composition of dietary carbohydrates can be designed so that they improve the glycemic and insulinaemic responses and increase satiety feeling. This can be detected in metabolic parameters in subjects with Mets.

The aim of our study is in subjects with Mets to compare the effect of acute consumption of bread rich in (a) purified AX, (b) purified BG, (c) rye bread with whole kernels (RK), with a (d) control group with consumption of white bread (WB).

The primary endpoint is GI. Secondary endpoints are the following items: glycemic load, insulin index, glucose, insulin, glucagon, inflammatory markers, incretins, rate of gastric emptying, and metabolomics. Also satiety feeling will be measured.

This project will improve opportunities for identifying and designing foods with low GI that is particularly suited to people who are at high risk of developing T2DM. The investigators also expect to gain a greater understanding of the metabolic fingerprint, as seen after ingestion of low-GI foods and thereby gain a molecular understanding of how low-GI foods affect health by altering metabolic processes. This will give us a deeper insight into the metabolic processes that are necessary for maintaining normal glucose homeostasis.

DETAILED DESCRIPTION:
Using a cross-over design, 12 subjects with Mets will consume test meals containing the four different bread types. Blood samples will be collected over 4,5 hours after ingestion of test meals containing around 145 g of each bread type, equivalent to 50 g available carbohydrate and 3 dl + 2 dl water on four different days in randomized order. Visual Analog Scale (VAS) will be used for determination of subjective satiety feeling and a subsequent meal will be served to estimate prospective food consumption.

ELIGIBILITY:
Inclusion Criteria:

* central obesity (Female > 94 cm; Male > 80 cm) with two of the following: -- fasting triglyceride (> 1,7 mmol/L)

  * HDL-cholesterol: (Female: < 1,03 mmol/L; Male: < 1,29 mmol/L)
  * blood pressure (≥ 130/85 mmHg)
  * fasting plasma glucose (≥ 5,6 mmol/L)) Subjects who are in medical treatment with lipid and blood pressure-lowering drugs can continue with their habitual treatment provided that the treatment is stable throughout the trial.

Exclusion Criteria:

* fasting plasma glucose > 7,0 mmol/l
* fasting plasma triglyceride > 5,0 mmol/l
* blood pressure > 160/100 mmHg
* legal incapacity
* endocrine, cardiovascular or kidney disease
* BMI > 38kg/m2
* corticosteroid treatment
* alcohol or drug addiction
* pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Glycaemic index of breads with arabinoxylan and beta-glucan compared with whole grain breads in subject with the metabolic syndrome | 4,5 hours

SECONDARY OUTCOMES:
Glycemic response and satiety | 4,5 hours
  glycemic load, insulin index, glucose, insulin, incretins, inflammatory markers, rate of gastric emptying, metabolomics, and satiety feeling

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Krishnan S, Hendriks HF, Hartvigsen ML, de Graaf AA. Feed-forward neural network model for hunger and satiety related VAS score prediction. Theor Biol Med Model. 2016 Jul 7;13(1):17. doi: 10.1186/s12976-016-0043-4. PMID 27387922
- [Derived] Nielsen KL, Hartvigsen ML, Hedemann MS, Laerke HN, Hermansen K, Bach Knudsen KE. Similar metabolic responses in pigs and humans to breads with different contents and compositions of dietary fibers: a metabolomics study. Am J Clin Nutr. 2014 Apr;99(4):941-9. doi: 10.3945/ajcn.113.074724. Epub 2014 Jan 29. PMID 24477039